CLINICAL TRIAL: NCT03654183
Title: Predictive Value of Intraoperative Indocyanine Green Clearance Test After Partially Blood Flow Blocking in Postoperative Liver Reserve: a Prospective Study
Brief Title: Predictive Value of Intraoperative Indocyanine Green Clearance Test After Partially Blood Flow Blocking in Postoperative Liver Reserve
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Lu Wang, MD, PhD, Head of Liver Surgery Department, Fudan University
Other Study IDs: LSD-2017-1-ICG
Record Dates: First submitted 2018-08-28; First posted 2018-08-31 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Predictive Value of ICG Clearance Measurement During Selective Hepatic Vascular Trial Clamping on Remnant Liver Function After Anatomic Liver Resection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Indocynine green clearance test — Indocyanine green clearance was determined by non-invasive pulse spectrophotometry (NIHON KOHDEN™; Pulse Dye Densito-Graph Analyzer, Japan).

SUMMARY:
Predictive value of intraoperative indocyanine green clearance measurement during selective hepatic vascular trial clamping on remnant liver function after anatomic liver resection.

DETAILED DESCRIPTION:
In this study, we will prospectively and consecutively enroll patients undergoing hemi-hepatectomy or lateral segmentectomy. ICG clearance measurements will be performed both preoperatively and intraoperatively under partial blood blocking of resecting segments. This study will use PHLF, C-D grade, MELD grade and postoperative hospital stay to evaluate and compare the potential of these measurements to predict postoperative liver function. Accordingly, we are supposed to demonstrate the sensitivity and specificity of intraoperative ICG clearance measurement in detecting postoperative liver failure. Furthermore, cut-off values would be defined to identify high, medium or low risk patients.

ELIGIBILITY:
Inclusion Criteria:

* (a) patients scheduled to undergo major anatomic liver resection according to clinical assessment, (b) patients'expectation of life longer than 3 months, and (c) age between 18 to 80 years old.

Exclusion Criteria:

* (a) patients could not tolerate liver surgery according to preoperative tests, (b) with no need for major liver resection according to intraoperative assessment, (c) had any contraindications to liver surgery, or (d) ICG metabolic disorder.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: (a) patients scheduled to undergo major anatomic liver resection according to clinical assessment, (b) patients'expectation of life longer than 3 months, and (c) age between 18 to 80 years old.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-08-31 (Estimated); Study Completion 2019-08-31 (Estimated)

PRIMARY OUTCOMES:
PHLF | 5 days after surgery
  Severe posthepatectomy liver failure (PHLF) was defined as Serum total bilirubin more than 120umol/L, prothrombin activity more than 50% or PHLF grade B/C. PHLF grade was defined by the International Study Group of Liver Surgery (ISGLS). Grade A PHLF requires no change of the patient's clinical management. The clinical management of patients with grade B PHLF deviates from the regular course but does not require invasive therapy. The need for invasive treatment defines grade C PHLF.
MELD score | 5 days after surgery
  The equation for the model for end-stage liver disease (MELD) score = 3.8×loge(bilirubin [mg/dL])+11.2×loge(INR)+9.6×loge(creatinine [mg/dL])+6.4×(etiology: 0 if cholestatic or alcoholic, 1 otherwise)
Clavien-Dindo grade | 5 days after surgery
  Grade I surgical complication was defined as any deviation from the normal postoperative course without the need for pharmacological treatment of surgical, endoscopic, and radiological interventions; grade II surgical complication was defined as requiring pharmacological treatment with drugs other than such allowed for grade I complications, blood transfusions and total parenteral nutrition are also included; grade III surgical complication was defined as requiring surgical, endoscopic or radiological intervention; grade IV surgical complication was defined as life-threatening complication requiring IC/ICU management; and grade V surgical complication was defined as death of a patient.

CONTACTS AND LOCATIONS:
Overall Officials: Lu Wang, MD, Study Director — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China